CLINICAL TRIAL: NCT03488485
Title: Efficacy of Decentralized Care in the Management of Patients With Hepatitis C in a Public Health Care Setting: The Punjab Model
Brief Title: Management of Patients With Hepatitis C in a Public Health Care Setting: The Punjab Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Directorate of Health and Family Welfare, Punjab (Other)
Responsible Party: Principal Investigator, Radha K Dhiman, Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IEC/2018/000324
Record Dates: First submitted 2018-03-22; First posted 2018-04-05 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Chronic Hepatitis c
Keywords: Mukh Mantri Punjab Hepatitis C Relief Fund,MMPHCRF; Direct antivirals, DAAs; Chronic hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Sofosbuvir; daclatasvir; ledipasvir

STUDY DESIGN:
Intervention Model Description: Real Life Efficacy Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DAA arm (Other): Direct Acting Antivirals therapy An algorithm was developed using DAA (Sofosbuvir-based regimens to treat all patients (RKD).
  Non Cirrhotics: Sofosbuvir (SOF)+ Daclatasvir (DCV) for 12-weeks
  Cirrhotics:
  Genotype 3 were treated with SOF+DCV+ ribavirin (RBV) for 24 weeks, Non-Genotype 3 patients were treated with SOF+LDV+RBV for 12-weeks or with SOF+LDV for 24-weeks (in RBV intolerant patients).
  Interventions: Drug: Direct Acting Antivirals

INTERVENTIONS:
Drug: Direct Acting Antivirals — DAAs given in patients with viremic chronic hepatitis C
  Other Names: Sofosbuvir; Daclatasvir; Ledipasvir

SUMMARY:
Background and Aims: The prevalence of hepatitis C virus infection (HCV) infection in Punjab, India is 3.29%, with an estimated burden of around 650,000 viremic chronic HCV (CHC) patients. The Mukh Mantri Punjab Hepatitis C Relief Fund (MMPHCRF) was launched in June 2016 to provide free treatment to all CHC aiming to eliminate HCV from Punjab. The study assessed the feasibility of decentralized care and efficacy and safety of 12 or 24 weeks of sofosbuvir (SOF) + ledipasvir (LDV) or SOF + daclatasvir (DCV) ± ribavirin (RBV) in the treatment of CHC patients in a public health care setting.

DETAILED DESCRIPTION:
An algorithm was developed using SOF-based regimens to treat all patients (RKD). Genotyping is not recommended for patients without cirrhosis of liver and they are being treated with SOF+DCV for 12-weeks, while genotyping is recommended for patients with cirrhosis of liver (Figure 1). Patients with liver cirrhosis and genotype 3 are being treated with SOF+DCV+RBV for 24 weeks, while non-genotype 3 patients are being treated with SOF+LDV+RBV for 12-weeks or with SOF+LDV for 24-weeks (in RBV intolerant patients). SVR-12 is mandatory in all patients. Methods: Decentralized care: All patients are being evaluated and treated at 3 Government Medical Colleges and 22 District Hospitals; they were followed up to 12 weeks post-treatment to look for sustained viral response (SVR-12). Health care worker capacity building: 90 medical specialists were trained in a 4-hr predefined course, followed by online continued medical education sessions by regular Extension for Community Healthcare Outcomes (ECHO) Clinic are being conducted fortnightly. 50 pharmacists, 2 from each of the 25 centres, dispense medicine as per specialist prescription. Data Management: 25 trained data entry operators and Clinton Health Access Initiative (CHAI) are managing epidemiological data on CHC hotspots, high-risk groups, local service providers, etc. Monitoring: Medical alerts are being used for compliance monitoring. Study design: A cost-effective algorithm has been developed using SOF-based regimens to treat all patients. The diagnosis of cirrhosis is based on clinical evidence including Aspartate Transaminase (AST)-to-platelet ratio index (APRI ≥ 2.0) and FIB-4 score (>3.25) or on liver stiffness measurement (LSM) ≥12.5 kilopascal (kPa) on fibroscan. The study aims to validate the efficacy and safety of generic all oral Direct Acting Antiviral (DAA) regimens in a decentralized algorithm based public health model in Punjab, India regardless of genotype/presence of cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Hepatitis C
* Age: >18 years

Exclusion Criteria:

* Chronic liver disease of a non-HCV etiology
* Serum Creatinine >1.5 mg/dl
* Evidence of hepatocellular carcinoma or other malignancy
* Significant cardiovascular, pulmonary, or neurological disease
* History of solid organ or bone marrow transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50000 (Estimated)
Dates: Start 2016-06-18 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Sustained Virological Response | Up to study completion ( average 12 -24 weeks after therapy)
  HCV RNA Load undetectable

SECONDARY OUTCOMES:
Serious adverse effects | Up to study completion ( average 12 -24 weeks after therapy)
  Assessment of drug related adverse effects, clinical events, decompensation of liver disease

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Premkumar M, Gupta E, Sandhu A, Sharma P, Nain J, Taneja S, Verma N, De A, Duseja A, Grover GS, Dhiman RK. Impact of Resistance Associated Substitutions and Predictors of Treatment Failure Following Direct-acting Antiviral Therapy in a Viral Hepatitis C Elimination Cohort. J Clin Exp Hepatol. 2025 Nov-Dec;15(6):102601. doi: 10.1016/j.jceh.2025.102601. Epub 2025 May 28. PMID 40611935
- [Derived] Premkumar M, Dhiman RK, Duseja A, Mehtani R, Taneja S, Gupta E, Gupta P, Sandhu A, Sharma P, Rathi S, Verma N, Kulkarni AV, Bhujade H, Chaluvashetty SB, Kalra N, Grover GS, Nain J, Reddy KR. Recompensation of Chronic Hepatitis C-Related Decompensated Cirrhosis Following Direct-Acting Antiviral Therapy: Prospective Cohort Study From a Hepatitis C Virus Elimination Program. Gastroenterology. 2024 Dec;167(7):1429-1445. doi: 10.1053/j.gastro.2024.08.018. Epub 2024 Aug 23. PMID 39181168